CLINICAL TRIAL: NCT03594929
Title: Effect of Remote Ischaemic preConditioning on Liver Injury in Patients Undergoing LIVER Resection Surgery: The ERIC-LIVER Trial
Brief Title: Effect of Remote Ischaemic preConditioning on Liver Injury in Patients Undergoing LIVER Resection Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The ERIC-LIVER trial
Record Dates: First submitted 2018-04-19; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active RIC (Active Comparator): Active RIC using a manual BP cuff to inflate to 200mmHg.
  Interventions: Device: Active RIC
- Sham Control (Sham Comparator): A sham control using a manual blood pressure cuff visually identical to that used in the RIC protocol will be placed on the upper arm and a simulated RIC protocol will be administered.
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Active RIC
  Arms: Active RIC
Device: Sham Control
  Arms: Sham Control

SUMMARY:
Liver resection has improved health outcomes in patients with hepatocellular carcinoma (HCC) in Singapore and worldwide. However, due to acute ischaemia/reperfusion injury (IRI) to the liver at the time of surgery, patients still experience significant morbidity and mortality. Therefore, novel therapies are required to protect the liver against acute IRI during partial hepatectomy. Remote ischaemic conditioning (RIC) using transient limb ischaemia/reperfusion has been shown to protect the liver in experimental animal studies. In the ERIC-LIVER trial the investigators investigate whether RIC can reduce liver injury and preserve liver function in patients with HCC undergoing partial hepatectomy.

DETAILED DESCRIPTION:
Liver resection has improved health outcomes in patients with hepatocellular carcinoma (HCC) in Singapore and worldwide. However, due to acute ischaemia/reperfusion injury (IRI) to the liver at the time of surgery, patients still experience significant morbidity and mortality. Therefore, novel therapies are required to protect the liver against acute IRI during partial hepatectomy. Remote ischaemic conditioning (RIC) using transient limb ischaemia/reperfusion has been shown to protect the liver in experimental animal studies. In the ERIC-LIVER trial the investigators investigate whether RIC can reduce liver injury and preserve liver function in patients with HCC undergoing partial hepatectomy.

50 patients with HCC undergoing partial hepatectomy will be randomised to receive either RIC (four-5 minute arm cuff inflations/deflations) or sham control (four-5 minute arm cuff simulated inflations/deflations) after induction of anesthesia and prior to surgical incision. The primary endpoint of the study will be acute liver injury assessed by serum transaminases measured at 24 hours post-resection. Secondary endpoints will include liver function in subset of patients (N=24, assessed by indocyanine green [ICG] clearance measured at 24 hours post-resection), incid ence of liver failure, episodes of confirmed sepsis, acute kidney injury, intensive care unit and hospital stay, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years and above
* Patients undergoing partial hepatectomy for primary HC

Exclusion Criteria:

* Patients with significant pulmonary disease (FEV1<40% predicted).
* Patients with known severe renal failure with a GFR<30 mL/min/1.73 m2.
* Patients on sulphonylurea or nicorandil, as these medications may interfere with the protective effect of RIC.
* Patients recruited into another study which may impact on this study. Significant peripheral arterial disease affecting the upper limbs.
* Patients undergoing repeat liver resection surgery.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08-15 (Actual); Primary Completion 2019-01-18 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
serum ALT (unit/L) following liver resection, measured at 24 hours | 24 hours
  serum ALT as a measure of acute liver injury
serum AST (unit/L) following liver resection, measured at 24 hours | 24 hours
  serum AST as a measure of acute liver injury

SECONDARY OUTCOMES:
serum ALT (unit/L) following liver resection, measured at 6 hours | 6 hours
  serum ALT as a measure of acute liver injury
serum ALT (unit/L) following liver resection, measured at 48 hours | 48 hours
  serum ALT as a measure of acute liver injury
serum ALT (unit/L) following liver resection, measured at 2 weeks | 2 weeks
  serum ALT as a measure of acute liver injury
serum AST (unit/L) following liver resection, measured at 6 hours | 6 hours
  serum AST as a measure of acute liver injury
serum AST (unit/L) following liver resection, measured at 48 hours | 48 hours
  serum AST as a measure of acute liver injury
serum ALT (unit/L) following liver resection, measured at 2 weeks | 2 weeks
  serum AST as a measure of acute liver injury
Indocyanine Green (ICG) retention test. | baseline in pre-admission clinic and post-operation day 1.
  Liver function as assessed by the ICG retention test. Testing is optional
Acute liver ischemia reperfusion injury on histology | up to 2 weeks
  Assessed by checking liver histology of the resected specimen
presence/absence of liver failure based on serum bilirubin and INR on post op day 5 | Baseline and day 5 post-surgery
  serum bilirubin and INR on post op day 5
Episodes of culture-confirmed sepsis | 30 days
  Episodes of culture-confirmed sepsis
Serum creatine (umol/L) | 3 days
  Measure of acute kidney injury based on rise in serum creatine on day 3 post op
ITU and hospital stay | Up to 30 days
  ITU and hospital stay
Rate of hospital admission | 30 days
  Rate of hospital admission
Mortality | 30 days
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided